CLINICAL TRIAL: NCT00002917
Title: A PHASE I/II INSTITUTIONAL STUDY OF INTRAVESICAL TAXOL (PACLITAXEL) INSTILLATION FOR THE TREATMENT OF SUPERFICIAL BLADDER CANCER
Brief Title: Paclitaxel in Treating Patients With Early-Stage Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mary Babb Randolph Cancer Center at West Virginia University Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: WVU-13707-OSP-97-092; CDR0000065299 (Registry Identifier: PDQ (Physician Data Query)); NCI-V97-1114
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2001-01

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of paclitaxel in treating patients with early-stage bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate toxicity and safety of intravesical paclitaxel in patients with superficial bladder cancer. II. Evaluate the efficacy of paclitaxel against transitional cell carcinoma in situ (CIS) and/or unresectable papillary superficial bladder cancer. III. Evaluate a dose-response effect and choose an appropriate dose for further clinical study.

OUTLINE: Cohorts of patients receive intravesical paclitaxel in escalating doses, administered twice weekly for 6 weeks, then once every 2 weeks for another 6 weeks, for a maximum of 2 courses at a dose level. Patients must complete 8 of the first 15 instillations and a 3 month cystoscopic exam with biopsy and cytology to be deemed evaluable. Participants are followed by quarterly cytoscopy and cytology for an additional 21 month period. Biopsies are performed at 3 and/or 6 months, and thereafter if clinically applicable.

PROJECTED ACCRUAL: 19 evaluable patients will be enrolled.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven CIS and/or unresectable/residual superficial bladder tumor (pTa G1-G3 to pT1 G1-G3) -confirmed by biopsy, bladder mapping, or positive cytology Cystoscopic examination and bladder mapping must be performed within 6 weeks of study

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: Karnofsky of 60 to 100% Life Expectancy: Not specified Hematopoietic: Hemoglobin greater than 11 g/dL WBC greater than 4500/mm3 Neutrophils greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin, AST, and ALT no greater than 2.5 x normal Renal: Creatinine no greater than 2.5 x normal Cardiovascular: No concurrent cardiovascular disease Other: No active infection requiring concurrent therapy Not pregnant or nursing No upper renal tract disease No concurrent malignancy except for basal or squamous cell skin cancer or noninvasive cancer of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No intravesical BCG within 3 months prior to study entry Prior BCG therapy is required for CIS patients (if not contraindicated) Chemotherapy: No prior intravesical chemotherapy within 4 weeks prior to study No prior systemic anticancer therapy within 4 months prior to study No prior paclitaxel therapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy within 4 months prior to study Surgery: Not specified Other: No hypersensitivity reactions to products containing cremophor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-11; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Lamm, MD, Study Chair — Mayo Clinic
Locations (1):
- West Virginia University Hospitals, Morgantown, West Virginia, United States